CLINICAL TRIAL: NCT00063531
Title: Coronary Disease Detection by Thallium SPECT and Fast CT
Brief Title: Comparison of Two Methods to Diagnose Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NA_00042276; R01HL071025 (NIH)
Record Dates: First submitted 2003-06-30; First posted 2003-07-01 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GeneSTAR participant meeting entry criteria: Healthy siblings of patients with early onset CAD (<60 years old) and the adult offspring of the siblings or probands

SUMMARY:
The purpose of this study is to compare two methods of diagnosing coronary artery disease (CAD), thallium single photon emission computed tomography (SPECT) and ultrafast computed tomography (CT).

DETAILED DESCRIPTION:
BACKGROUND:

The ability to noninvasively detect CAD at a subclinical stage is fundamental to understanding the biology of the transition of occult CAD to clinical CAD in asymptomatic people at the highest risk for future CAD.

DESIGN NARRATIVE:

The cross-sectional study is designed to identify the factors explaining why some individuals have exercise ischemia without significant coronary artery calcium (CAC) while others have extensive CAC without exercise ischemia. The investigators will compare the pathophysiological features of a functional test for subclinical CAD detection (exercise radionuclide perfusion SPECT) and an anatomical test to detect coronary calcification (ultrafast CT) in a high-risk asymptomatic population of 30 to 59 year old siblings of people with premature CAD. Siblings will undergo screening for occult CAD using both detection methods. Individuals who are abnormal on either test (exercise-induced ischemia or calcium score greater than 75th percentile for age and sex) will be offered cardiac catheterization, which will include quantitative coronary angiography, assessment of endothelial function by intracoronary acetylcholine, and measurement of plaque volume and composition in a selected coronary artery by intravascular ultrasound (IVUS). The study will focus on the pathophysiology of occult CAD among individuals who have exercise ischemia with low calcium scores and other individuals who have high calcium scores without ischemia. Discrepancies between these two tests measure potentially different biological pathways and such discrepancies are observed frequently in high-risk asymptomatic siblings (40% in our recent pilot study). Analyses will be done to determine which biological risk factors can account for variation in plaque calcification that results in discordances between these two measures of occult disease (including lipid levels and subclasses, Lp(a), diabetes, thrombotic factors, pro-inflammatory cytokines, and importantly, those factors involved in calcium regulation, and bone regulatory proteins). In those siblings undergoing cardiac catheterization, analyses will be done to determine whether the severity or extent of coronary luminal narrowing, the presence of epicardial or microvascular endothelial dysfunction, or the volume or calcium content of plaque by IVUS can account for discordances between the two screening tests. Polymorphisms in several candidate genes that may affect tissue calcification will be examined as a possible explanation for variations in plaque calcification as reflected in test discordance. Plasma and DNA will also be collected for novel studies of factors that may account for variability in coronary plaque calcification in this unique well characterized asymptomatic high risk population. This will be the first comprehensive study to define the unique biological and genetic factors related to occult CAD, as detected by both perfusion imaging and ultrafast CT.

ELIGIBILITY:
Inclusion Criteria:

* Siblings of hospitalized index patients with documented CAD prior to 60 years of age
* Index patients who have demonstrated angiographic lesions greater than or equal to 50% in greater than or equal to 1 vessel, accompanied by angina or a documented CAD event
* Siblings with no known history of CAD
* Siblings with a positive screening test for occult CAD (abnormal ETT or thallium scan, or CAC score greater than 75th percentile) will be invited for coronary angiography

Exclusion Criteria:

* Index patients with CAD associated with some other primary disease (e.g., collagen vascular disease, transplantation, or chronic corticosteroid therapy)
* Siblings with a life-threatening comorbidity (e.g., AIDS, cancer)
* Siblings who have had an organ transplant
* Siblings receiving chronic glucocorticosteroids
* Siblings with known collagen vascular disease
* Siblings with a limitation that would preclude the capacity to exercise sufficiently for the test
* Siblings unable to give informed consent

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy siblings of patients with early onset CAD (<age 60) or the adult offspring of the siblings or probands, all participants in the GeneSTAR study.
Sampling Method: Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2003-06; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity of CAC vs coronary plaque volume for detecting CAD by CTA | Concurrent with CTA
  The question to be answered is what percentage of healthy people with a family history of early onset CAD in a sibling have only non-calcified coronary artery plaque that would not be detected by coronary calcium imaging. How much additional information is provided by CTA?

CONTACTS AND LOCATIONS:
Overall Officials: Lewis C. Becker, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States